CLINICAL TRIAL: NCT01170702
Title: The Postoperative Analgesic Efficacy of Varied Concentrations of Ropivacaine Used for the Transverse Abdominis Plane (TAP) Block After Cesarean Delivery
Brief Title: Transverse Abdominis Plane (TAP) Block After Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Walega, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00008429
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Results first posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Postoperative Pain; Pregnancy; Obesity
Keywords: Cesarean Delivery; Ropivicaine; TAP block
MeSH Terms: conditions — Pain, Postoperative; Obesity | interventions — Saline Solution; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Placebo Comparator): TAP Block utilizing 15mL of 0.9% normal saline per side
  Interventions: Drug: 0.9% Normal Saline
- Group 2 (Experimental): TAP Block utilizing 15ml of 0.2% ropivacaine per side
  Interventions: Drug: 0.2% Ropivacaine
- Group 3 (Experimental): TAP Block utilizing 15ml of 0.5% ropivacaine per side
  Interventions: Drug: 0.5% Ropivacaine
- Group 4 (Experimental): TAP Block utilizing 15ml of 0.75% ropivacaine per side
  Interventions: Drug: 0.75% Ropivacaine

INTERVENTIONS:
Drug: 0.9% Normal Saline — The abdominal muscle layers will be located by placing the ultrasound transducer perpendicular to the coronal anatomic plane at the T-10 dermatome level in the patient's midaxillary line. Under ultrasound guidance, a 70mm or 90mm, 21 gauge blunted Stimuplex needle will be advanced from the skin until the tip reaches the fascial layer between the internal oblique and transversus abdominis. 15ml of the study drug will be injected incrementally. The needle will then be removed and the process repeated in the same manner on the patient's opposite side.
  Arms: Group 1
Drug: 0.2% Ropivacaine — The abdominal muscle layers will be located by placing the ultrasound transducer perpendicular to the coronal anatomic plane at the T-10 dermatome level in the patient's midaxillary line. Under ultrasound guidance, a 70mm or 90mm, 21 gauge blunted Stimuplex needle will be advanced from the skin until the tip reaches the fascial layer between the internal oblique and transversus abdominis. 15ml of the study drug will be injected incrementally. The needle will then be removed and the process repeated in the same manner on the patient's opposite side.
  Arms: Group 2
Drug: 0.5% Ropivacaine — The abdominal muscle layers will be located by placing the ultrasound transducer perpendicular to the coronal anatomic plane at the T-10 dermatome level in the patient's midaxillary line. Under ultrasound guidance, a 70mm or 90mm, 21 gauge blunted Stimuplex needle will be advanced from the skin until the tip reaches the fascial layer between the internal oblique and transversus abdominis. 15ml of the study drug will be injected incrementally. The needle will then be removed and the process repeated in the same manner on the patient's opposite side.
  Arms: Group 3
Drug: 0.75% Ropivacaine — The abdominal muscle layers will be located by placing the ultrasound transducer perpendicular to the coronal anatomic plane at the T-10 dermatome level in the patient's midaxillary line. Under ultrasound guidance, a 70mm or 90mm, 21 gauge blunted Stimuplex needle will be advanced from the skin until the tip reaches the fascial layer between the internal oblique and transversus abdominis. 15ml of the study drug will be injected incrementally. The needle will then be removed and the process repeated in the same manner on the patient's opposite side.
  Arms: Group 4

SUMMARY:
Since there have been no published dose-response studies investigating the effective analgesic dose of ropivacaine for use in a TAP block for post-Cesarean delivery analgesia, the investigators propose a study primarily examining the effect on 24 hour post-Cesarean delivery opioid consumption of using either a placebo, 0.25% ropivacaine, 0.5% ropivacaine, or 0.75% ropivacaine for TAP blocks.

DETAILED DESCRIPTION:
Cesarean delivery is the most commonly performed surgical procedure in the United States today, with over 1.2 million cases performed in 2005. One of the most important aspects of cesarean delivery is the provision of safe, effective postoperative analgesia for the mother, while simultaneously ensuring minimal side effects for both the mother and neonate. Studies have suggested that a multimodal approach to post-cesarean pain utilizing both intravenous, oral, and neuraxial opioids and non-steroidal anti-inflammatory drugs is highly effective in providing effective analgesia.

A significant component of post-cesarean pain is incisional pain from the Pfannenstiel incision on the anterior abdominal wall. The sensory supply to the skin, muscles, and parietal peritoneum of the anterior abdominal wall is derived from the anterior rami of T7-L1. After exiting the spinal column, these nerves proceed through the lateral abdominal wall within the transversus abdominal fascial plane, terminating in the anterior abdominal wall.

Recent studies have suggested that blocking these afferent sensory nerves with local anesthetics, as part of a multimodal postoperative pain regimen, provides superior pain relief in terms of decreased pain scores and morphine consumption for up to 48 hours postoperatively. The technique utilized for these studies employed a surface anatomical approach to the transversus abdominal fascial plane via the lumbar triangle of Petit, a technique validated in both cadaveric and radiologic studies. However, as ultrasonography has emerged as the "gold standard" for initiating many nerve blocks, reports have described the successful use of ultrasound imaging for initiation of transversus abdominis plane (TAP) blocks for both abdominal surgeries and cesarean deliveries.

In the published studies investigating the use of the TAP block for post-operative analgesia, either ropivacaine or bupivacaine was utilized in concentrations of 0.75% and 0.375%, respectively. Studies comparing ropivacaine with bupivacaine for use in interscalene, femoral, or sciatic nerve blocks have found no difference in terms of potency, time to onset or duration of postoperative analgesia between the two local anesthetics. Although no similar studies have been done with TAP blocks, one can assume that utilization of ropivacaine for this nerve block would yield similar results in terms postoperative analgesia. Moreover, the cardiotoxicity of ropivacaine has been shown to be significantly less than bupivacaine, making it a safer alternative for use in nerve blocks when used in high doses.

Risk factors for respiratory depression after the administration of neuraxial opioids in the non-obstetric population include morbid obesity and obstructive sleep apnea. For the obstetric population, a study of 856 patients revealed that all 8 patients who experienced respiratory depression after intrathecal morphine for cesarean delivery were markedly obese. Furthermore, the onset of respiratory depression after intrathecal morphine can occur up to 12 hours after administration, a time period when the patient is not being as closely monitored as she is during the 1:1 nursing care in the recovery room. Therefore, it is the investigators policy on the Labor and Delivery unit to not administer intrathecal morphine to any parturient with a history of obstructive sleep apnea or a BMI > 40 kg/m2. These patients often require intravenous opioid patient-controlled analgesia postoperatively, which has been shown to provide inferior pain relief and greater opioid consumption than neuraxial opioids. The current clinical standard is to administer the TAP block to those patients who have not received morphine in their neuraxial anesthetic. The TAP block offers a novel addition to the management of post-cesarean pain for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* ASA II-III patient
* > 18 years of age who is pregnant
* presenting for a cesarean delivery via Pfannenstiel incision who is eligible to receive a spinal anesthetic with 0.75% bupivacaine and fentanyl and whose is not eligible to receive intrathecal morphine due to a BMI >40 kg/m2.

Exclusion Criteria:

* < 18 years of age
* contraindication to placement of a spinal anesthetic
* contraindication to use of non-steroidal anti-inflammatory drugs (NSAIDs)
* patients receiving medical therapies considered to result in tolerance to opioids
* patients with a history of established chronic pain, (e.g. chronic low back pain, fibromyalgia or headaches), defined as requiring regular medical follow-up with pain specialists, as well as recent use (within the year preceding pregnancy) of opioid analgesics as an outpatient
* patients with a history of diabetes mellitus
* patients undergoing a vertical midline skin incision
* patients who are undergoing a cesarean delivery after a failed vaginal trial of labor
* patients who had a prior epidural placed for labor analgesia during the same hospital encounter.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Walega, M.D., Study Director — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardoso MM, Carvalho JC, Amaro AR, Prado AA, Cappelli EL. Small doses of intrathecal morphine combined with systemic diclofenac for postoperative pain control after cesarean delivery. Anesth Analg. 1998 Mar;86(3):538-41. doi: 10.1097/00000539-199803000-00017. PMID 9495409
- [Background] Lowder JL, Shackelford DP, Holbert D, Beste TM. A randomized, controlled trial to compare ketorolac tromethamine versus placebo after cesarean section to reduce pain and narcotic usage. Am J Obstet Gynecol. 2003 Dec;189(6):1559-62; discussion 1562. doi: 10.1016/j.ajog.2003.08.014. PMID 14710063
- [Background] Siddik SM, Aouad MT, Jalbout MI, Rizk LB, Kamar GH, Baraka AS. Diclofenac and/or propacetamol for postoperative pain management after cesarean delivery in patients receiving patient controlled analgesia morphine. Reg Anesth Pain Med. 2001 Jul-Aug;26(4):310-5. doi: 10.1053/rapm.2001.21828. PMID 11464348
- [Background] Loos MJ, Scheltinga MR, Mulders LG, Roumen RM. The Pfannenstiel incision as a source of chronic pain. Obstet Gynecol. 2008 Apr;111(4):839-46. doi: 10.1097/AOG.0b013e31816a4efa. PMID 18378742
- [Background] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] O'Donnell BD, McDonnell JG, McShane AJ. The transversus abdominis plane (TAP) block in open retropubic prostatectomy. Reg Anesth Pain Med. 2006 Jan-Feb;31(1):91. doi: 10.1016/j.rapm.2005.10.006. No abstract available. PMID 16418039
- [Background] Walter EJ, Smith P, Albertyn R, Uncles DR. Ultrasound imaging for transversus abdominis blocks. Anaesthesia. 2008 Feb;63(2):211. doi: 10.1111/j.1365-2044.2007.05424.x. No abstract available. PMID 18211466

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 120 patients were randomized to one of four groups who received TAP blockade. Four patients subsequently were dropped from the study after randomization for pre-defined criteria. Substantive data was missing in one subject who was excluded from analysis. One patient received a morphine PCA instead of hydromorphone due to a drug shortage.
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 34 | 32 | 25 | 29
Completed | 33 | 30 | 25 | 27
Not Completed | 1 | 2 | 0 | 2
Not completed — Exclusion criteria met after consent | 1 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 34 | 32 | 25 | 29 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 32 | 25 | 29 | 120
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 25 | 29 | 120
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 32 | 25 | 29 | 120
BMI (kg/m^2) [Median (Full Range); unit: BMI (kg/m^2)] — The BMI is the subjects weight in kilograms (kg) divided by his or her height in meters squared.
  BMI (kg/m^2) | 44.3 [39 to 52] | 43.7 [40 to 51] | 44.6 [40 to 53] | 44.5 [41 to 53] | 44.28 [39 to 53]
Estimated Gestational Age (EGA) [Median (Inter-Quartile Range); unit: weeks] — Estimated gestational age in weeks.
  weeks | 39 [39 to 39] | 39 [38 to 39] | 39 [39 to 40] | 39 [38 to 39] | 39 [38 to 40]
# previous Cesarean deliveries [Count of Participants; unit: Participants] — Population: 1 subject did not respond for saline group previous cesarean delivery
  Participants
    number analyzed (Participants) | 33 | 30 | 25 | 27 | 115
    No Cesarean Deliveries | 12 | 9 | 12 | 9 | 42
    1 Cesarean Delivery | 21 | 14 | 11 | 12 | 58
    > 1 Cesarean Deliveries | 0 | 7 | 2 | 6 | 15
Race/Ethnicity [Count of Participants; unit: Participants]
  Race of Participants : Caucasian | 19 | 13 | 12 | 10 | 54
  Race of Participants : African American | 9 | 8 | 7 | 10 | 34
  Race of Participants : Asian | 1 | 1 | 1 | 0 | 3
  Race of Participants : Hispanic | 4 | 8 | 5 | 7 | 24
  Other | 1 | 2 | 0 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Morphine Equivalents 0-24 Hours (Mgs)
Description: Total dose of morphine equivalents (IV equivalent of morphine) taken by the participant 0-24 hours after completion of the TAP block.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: Morphine equivalents (mg)
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 34 | 32 | 25 | 29
Morphine equivalents (mg) | 54 [37 to 70] | 38 [22 to 46] | 32 [18 to 54] | 45 [29 to 75]
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3 vs Group 4; Test type: Non-Inferiority — The non inferiority margin is clinically important reduction in 24 hour hydromorphone consumption of 25%, 37.5% and 50% absolute reduction, compared with control; p = .05, Kruskal-Wallis; Median Difference (Final Values) = 1.25, .975% CI 2-sided [1.25 to 1.25], Standard Deviation .05

2. Secondary Outcome: Morphine Equivalents 24-72 Hours (Mgs)
Description: Total dose of morphine equivalents (IV equivalent of morphine) taken by the participant 24-72 hours after completion of the TAP block.
Time Frame: 24-72 hours
Measure: Median (Inter-Quartile Range); unit: Morphine equivalents (mgs)
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 34 | 32 | 25 | 29
Morphine equivalents (mgs) | 67 [50 to 73] | 60 [27 to 73] | 67 [60 to 80] | 67 [47 to 107]

3. Secondary Outcome: Morphine Equivalents Total (Mgs)
Description: Total dose of morphine equivalents (IV equivalent of morphine) taken by the participant 0-72 hours after completion of the TAP block.
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: Morphine equivalents (mgs)
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 34 | 32 | 25 | 29
Morphine equivalents (mgs) | 120 [90 to 158] | 96 [57 to 117] | 98 [82 to 129] | 112 [82 to 182]

4. Secondary Outcome: Time to First PCA Request
Description: The elapsed time in minutes of the first PCA (patient controlled analgesia) request in time (minutes) from the end of the TAP block.
Time Frame: Elapsed time in minutes
Measure: Mean (Inter-Quartile Range); unit: Minutes
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 34 | 32 | 25 | 29
Minutes | 90 [40 to 112] | 118 [69 to 157] | 126 [75 to 182] | 83 [41 to 143]

5. Secondary Outcome: Pain Scores at Rest
Description: Pain scores at rest ( 0 low 10 high) using an 11 point VRS (verbal pain scale) at the following hour time points, at the first request for patient controlled analgesia (PCA) then at 2,6,24,and 74 hours after the first request for PCA (patient controlled analgesia).
Time Frame: Request for first patient controlled analgesia then at 2,6,24,72 hours after initial PCA request
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 34 | 32 | 25 | 29
units on a scale
  At first PCA request | 3 [2 to 4.5] | 3 [0 to 3] | 2 [0 to 4] | 2 [1 to 4]
  2 hous after first PCA request | 3 [1 to 5] | 1 [0 to 3] | 0 [0 to 3] | 2 [0 to 3]
  6 hours after first PCA request | 3 [2 to 5] | 2 [1 to 3] | 2 [1 to 3] | 2 [0 to 4]
  24 hours after first PCA request | 2 [1 to 3] | 1 [0 to 2] | 1 [0 to 2] | 3 [1 to 4]
  72 hours after first PCA reqest | 1 [0 to 3] | .5 [0 to 1] | 1 [0 to 2] | 1 [0 to 4]

6. Secondary Outcome: Pain Scores With Movement
Description: Pain scores with movement ( 0 low 10 high) using an 11 point VRS (verbal pain scale) at the first request for patient controlled analgesia (PCA) then at 2,6,24,and 74 hours after the first request for PCA (patient controlled analgesia).
Time Frame: First PCA request then at 2,6,24,72 hours after first PCA request.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 34 | 32 | 25 | 29
units on a scale
  At first PCA request | 5 [3 to 6] | 3.5 [2 to 5] | 3.5 [1 to 7] | 4 [2 to 5]
  2 hous after first PCA request | 4 [1.5 to 5.5] | 2 [1 to 5] | 3 [1 to 6] | 3 [1 to 4]
  6 hours after first PCA request | 4 [3 to 6] | 4 [3 to 6] | 5 [4 to 6] | 4 [3 to 6]
  24 hours after first PCA request | 4 [3 to 5] | 3 [2 to 4] | 4 [2 to 5] | 5 [4 to 8]
  72 hours after first PCA reqest | 3.5 [2 to 5] | 2 [1 to 4] | 3 [2 to 4] | 4 [2 to 6]

7. Secondary Outcome: Pain Burden at Rest
Description: Pain burden at rest calculated as area under the pain score * time (hr) curve 0-72 hours.
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: score on scale * (hr)
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 34 | 32 | 25 | 29
score on scale * (hr) | 129 [84 to 195] | 79 [33 to 130] | 79 [48 to 133] | 151 [68 to 243]

8. Secondary Outcome: Pain Burden With Movement
Description: Pain burden with movement calculated as area under the pain score * time (hr) curve 0-72 hours.
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: pain score * time (hr) curve 72 hours
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 34 | 32 | 25 | 29
pain score * time (hr) curve 72 hours | 265 [221 to 320] | 202 [120 to 278] | 233 [202 to 289] | 327 [217 to 417]

ADVERSE EVENTS:
Time Frame: Two hours after TAP block
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32 | 0/25 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32 | 0/25 | 0/29
Other Adverse Events (participants affected / at risk) | 11/34 | 8/32 | 12/25 | 10/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=34) | Group 2 (N=32) | Group 3 (N=25) | Group 4 (N=29)
Nausea 2 hours after TAP (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (10) | 7 (7) | 12 (12) | 8 (8) — Pruritus 2 hours after TAP block

LIMITATIONS AND CAVEATS:
We did not evaluate TAP success by quantifying the area of cutaneous sensory blockade. We established baseline pain scores immediately prior to TAP blockade, although most blocks were performed with residual spinal blockade present.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT01170702/Prot_SAP_000.pdf